CLINICAL TRIAL: NCT07380750
Title: A Cluster Randomized Control Trial of a Family-Centered School Physical Activity Program to Improve Early Adolescent Mental Health in China
Brief Title: Active Families, Healthy Minds: A Family-Centered School Physical Activity Program for Early Adolescents
Acronym: AFHM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Ma Ruisi, Principal Investigator, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBRE-25-0397
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Adolescent Mental Health; Physical Inactivity; Mental Well-being; Sedentary Behavior
Keywords: Physical Activity; Family-based Intervention; School-based Intervention; Self-Determination Theory; Early Adolescence; Mental Health Promotion; Prevention
MeSH Terms: conditions — Sedentary Behavior; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial. Schools were the unit of randomization (clusters), assigned in a 1:1:1 ratio to the intervention, active control, or wait-list control arm.
Who Masked: Outcomes Assessor
Masking Description: Data analysts were also masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family-Supported Intervention (Experimental): Students participate in structured school-based physical activity sessions twice a week. Additionally, families implement weekly home activity routines (one weekday, one weekend) supported by goal-setting sheets and WeChat prompts to foster parental engagement.
  Interventions: Behavioral: Family-Supported PA Program
- Active Control (School-Only PA) (Active Comparator): Students participate in the same structured school-based physical activity sessions (twice a week) as the intervention group. They receive general health handouts but do not engage in structured family routines or receive home-based support.
  Interventions: Behavioral: School-Only PA Program
- Wait-List Control (Other): Students continue with the standard school curriculum and routine physical education classes. They receive no additional intervention during the study period but are offered educational materials after the final assessment.
  Interventions: Behavioral: Standard Physical Education

INTERVENTIONS:
Behavioral: Family-Supported PA Program — Consists of two components:
  School component: Structured aerobic games and skills practice delivered by PE teachers twice a week.
  Home component: Weekly parent-child joint activity routines (one weekday, one weekend) supported by goal-setting sheets. Parents receive weekly WeChat prompts to facilitate planning and positive communication.
  Arms: Family-Supported Intervention
Behavioral: School-Only PA Program — Consists of structured aerobic games and skills practice delivered by PE teachers twice a week (same frequency and intensity as the family intervention). Participants receive general health education handouts but do not engage in structured family routines or receive home-based support.
  Arms: Active Control (School-Only PA)
Behavioral: Standard Physical Education — Participants continue with the standard school curriculum and routine physical education classes. No additional structured activities or materials are provided during the study period.
  Arms: Wait-List Control

SUMMARY:
This study evaluates the effectiveness of a family-centered school physical activity program, titled "Active Families, Healthy Minds," designed to improve mental health among early adolescents (ages 10-14) in China.

In response to high academic pressure and low physical activity levels, this program integrates structured physical education sessions at school with simple, interactive home-based activity routines involving parents. The study compares this family-supported intervention against a standard school-only physical activity program and a wait-list control group. The primary goal is to determine if involving parents in school-based physical activity initiatives leads to better mental well-being, increased habitual physical activity, and stronger family support compared to school-only approaches.

DETAILED DESCRIPTION:
Adolescent mental health is a significant public health concern, particularly in China where academic pressure often limits opportunities for physical activity (PA). This cluster randomized controlled trial (RCT) tests a "Active Families, Healthy Minds" program built on Self-Determination Theory (SDT), targeting the satisfaction of basic psychological needs (autonomy, competence, and relatedness).

The study involves three parallel arms:

Intervention Group (Family-Supported Program): Students participate in structured aerobic games during school PE sessions (twice weekly). Additionally, families implement a home component consisting of one weekday and one weekend joint activity. Parents and children co-plan activities using goal sheets and receive weekly prompts via the WeChat app to facilitate planning and positive communication.

Active Control Group: Students receive the same dose of school-based physical activity (frequency, intensity, and content) as the intervention group but without the structured family engagement component or home routines.

Wait-list Control Group: Students continue with the standard school curriculum and routine services without additional intervention.

The primary outcome is mental well-being, measured by the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Secondary outcomes include basic psychological need satisfaction, habitual physical activity levels, physical literacy, exercise enjoyment, exercise motivation, and parental support. Data are collected at baseline and at 2, 4, and 6 months follow-up to assess the trajectory of change.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a student at the participating study schools.
* Aged between 10 and 14 years.
* Provided written parental consent and written student assent.
* Able to comprehend and complete questionnaires in Chinese.
* Judged by the school health team as safe to participate in moderate-intensity physical activity.

Exclusion Criteria:

* Having a physician-advised restriction on exercise.
* Suffering from an acute illness at the time of baseline assessment.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Mental Well-being (WEMWBS) | Baseline, 2 months, 4 months, and 6 months
  Assessed using the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). The scale contains 14 positively worded items rated on a 5-point Likert scale (from 1 = 'none of the time' to 5 = 'all of the time'). Total scores range from 14 to 70, with higher scores indicating better mental well-being.

SECONDARY OUTCOMES:
Basic Psychological Need Satisfaction (BPNS) | Baseline, 2 months, 4 months, and 6 months
  Assessed using a 21-item scale aligned with autonomy, competence, and relatedness. Higher scores reflect stronger satisfaction of psychological needs.
Habitual Physical Activity | Baseline, 2 months, 4 months, and 6 months
  A composite score derived from a weekly activity checklist and school day/weekend frequency items, aligned with the Physical Activity Questionnaire for adolescents. Higher scores indicate higher activity levels.
Physical Literacy (PPLI-SC) | Baseline, 2 months, 4 months, and 6 months
  Assessed using the Perceived Physical Literacy Instrument (Simplified Chinese version). It consists of 8 items rated on a 5-point Likert scale. Total scores range from 9 to 45, with higher scores reflecting higher perceived physical literacy.
Parental Support for Physical Activity | Baseline, 2 months, 4 months, and 6 months
  Assessed using items from the Activity Support Scale for Multiple Groups (ACTS-MG), measuring modeling, co-participation, transport, and monitoring. Separate scores for fathers and mothers. Higher scores indicate greater support.
Body Mass Index (BMI) | Baseline, 2 months, 4 months, and 6 months
  Calculated as weight in kilograms divided by height in meters squared (kg/m^2). Height and weight were measured by staff using calibrated equipment.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education, Jinan University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided